CLINICAL TRIAL: NCT03031418
Title: Clinical Evaluation of the 'ExoDx Prostate IntelliScore' in Men Presenting for Initial Biopsy; Additional Confirmation Study Including Impact on Decision-making and Health Economics.
Brief Title: Clinical Evaluation of the 'ExoDx Prostate IntelliScore' (EPI)
Status: Completed | Type: Observational
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2016-001
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Random first catch urine sample > 20mL
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Enroll up to 500 patients to confirm performance of ExoDx Prostate IntelliScore (EPI) for men scheduled for initial biopsy. The treating physician will collect a urine sample from from a consented subject to test before their scheduled prostate biopsy (during your established clinic visit).
- Cohort 2: Enroll up to 500 patients to evaluate how the results of the urine test influences the decision process for determining whether to perform a prostate biopsy. The treating physician will collect a urine sample for testing and 2 weeks later discuss whether to perform a prostate biopsy with the subject knowing the results of the urine test and comparing them to the overall consensus report from Cohort 1 as well as other clinical factors the treating physician would otherwise use to determine whether they should have a prostate biopsy.
  Interventions: Diagnostic Test: ExoDx Prostate Intelliscore

INTERVENTIONS:
Diagnostic Test: ExoDx Prostate Intelliscore — ExoDx Prostate (IntelliScore) is a non-invasive, urinary 3-gene expression validated test in which the results of the assay are adjunctive to the ordering physician's clinical judgment and work-up of the patient in the determination of whether a prostate needle biopsy is necessary. The ExoDx Prostate (IntelliScore) was clinically validated to discriminate patients with higher grade prostate cancer from those with more indolent lower grade cancer and benign disease.
  Other Names: EPI
  Groups: Cohort 2

SUMMARY:
The purpose of this research study is investigate a new and validated urine test which predicts the likelihood of high grade prostate cancer on an initial prostate biopsy The current protocol has two objectives; one is to further assess and evaluate the performance of the urine test in men already scheduled for initial prostate needle biopsy (cohort (group) 1) and two, to evaluate how the results of the urine test influences the decision process for determining whether to perform a prostate biopsy (cohort (group) 2).

DETAILED DESCRIPTION:
Primary Objective(s)

* Confirm performance of the ExoDx Prostate (IntelliScore) (EPI) utilizing a designated collection vessel for men presenting for their initial prostate biopsy with an elevated Prostate-specific antigen (2-10 ng/mL).
* Evaluate impact of the confirmed ExoDx Prostate (IntelliScore) on the decision to perform an initial prostate biopsy for men presenting with an elevated Prostate-specific antigen (2-10 ng/mL).

Secondary and Exploratory Objectives

* Assess physician satisfaction with the ExoIntelliScore Prostate report including test result presentation, graphics and interpretation.
* Assess patient satisfaction for ease of understanding test results and role on decision process to have a biopsy.
* Determine the medical economic impact of the ExoIntelliScore Prostate in the prostate biopsy decision process.
* Correlation of the ExoIntelliScore Prostate score with the actual biopsy result.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age
* Clinical suspicion for prostate cancer
* Elevated Prostate-specific antigen between: 2.0 - 10 ng/ mL
* No clinical history of a prior negative biopsy

Exclusion Criteria:

* History of prior prostate biopsy.
* Use of medications or hormones that are known to affect serum Prostate-specific antigen levels within 3-6 months of study enrollment.
* Clinical symptoms of urinary tract infection (including prostatitis) at the time of enrollment.
* History of prostate cancer.
* History of invasive treatments for benign prostatic hypertrophy (Benign Prostatic Hyperplasia) or lower urinary track symptoms within 6 months of study enrollment.
* No known hepatitis (all types) and/or HIV documented in patient's medical record.
* Patients with history of concurrent renal/bladder tumors.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be male to screen for prostate cancer
Study Population: Male, 50+ years of age with a clinical suspicion for prostate cancer based in part on an elevated Prostate-specific antigen (limit range: 2.0 - 10 ng/ mL), and or suspicious DRE, without the clinical history of a prior negative biopsy.
Sampling Method: Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Confirm performance of the ExoDx Prostate IntelliScore | 6 months
  Confirm performance of the ExoDx Prostate IntelliScore utilizing a designated collection vessel for men presenting for their initial prostate biopsy with an elevated prostate-specific antigen (2-10 ng/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Roger Tun, Study Director — Exosome Diagnostics, Inc.
Locations (18):
- United States (18):
  - 21st Century Oncology, Fort Myers, Florida
  - Mount Sinai Medical Center of Florida, Miami, Florida
  - Southeastern Urology Associates, Macon, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Walter Reed National Military Medical CPDR, Bethesda, Maryland
  - Comprehensive Urology, Royal Oak, Michigan
  - Five Valley Urology, Missoula, Montana
  - Premier Urology Group, Edison, New Jersey
  - Urologic Research and Consulting LLC, Englewood, New Jersey
  - Delaware Valley Urology, Voorhees Township, New Jersey
  - Manhattan Medical Research, New York, New York
  - NYU Urology Associates, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - UT Health Science Center, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Donovan MJ, Noerholm M, Bentink S, Belzer S, Skog J, O'Neill V, Cochran JS, Brown GA. A molecular signature of PCA3 and ERG exosomal RNA from non-DRE urine is predictive of initial prostate biopsy result. Prostate Cancer Prostatic Dis. 2015 Dec;18(4):370-5. doi: 10.1038/pcan.2015.40. Epub 2015 Sep 8. PMID 26345389
- [Derived] Kretschmer A, Tutrone R, Alter J, Berg E, Fischer C, Kumar S, Torkler P, Tadigotla V, Donovan M, Sant G, Skog J, Noerholm M. Pre-diagnosis urine exosomal RNA (ExoDx EPI score) is associated with post-prostatectomy pathology outcome. World J Urol. 2022 Apr;40(4):983-989. doi: 10.1007/s00345-022-03937-0. Epub 2022 Jan 27. PMID 35084544
- [Derived] McKiernan J, Donovan MJ, Margolis E, Partin A, Carter B, Brown G, Torkler P, Noerholm M, Skog J, Shore N, Andriole G, Thompson I, Carroll P. A Prospective Adaptive Utility Trial to Validate Performance of a Novel Urine Exosome Gene Expression Assay to Predict High-grade Prostate Cancer in Patients with Prostate-specific Antigen 2-10ng/ml at Initial Biopsy. Eur Urol. 2018 Dec;74(6):731-738. doi: 10.1016/j.eururo.2018.08.019. Epub 2018 Sep 17. PMID 30237023